CLINICAL TRIAL: NCT00694096
Title: Sunitinib for Metastatic Renal Cell Cancer With Imaging Biomarker Assessments for the Early Prediction of Tumor Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI21897
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-10

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Imaging studies with complete analyses will be provided on all patients prior to institution of sunitinib therapy as well as after therapy at various early time points (1 week in 5 patients, 2 weeks in 5 patients, 3 weeks in 5 patients or 4 weeks in 5 patients) after institution of sunitinib therapy at 37.5 mg orally/day.
  Imaging studies include:
  FDG-PET scans FLT-PET scans H215O-PET scans DCE-MRI scans
  Other Names: Sutent®

SUMMARY:
This exploratory clinical study is designed to obtain pre-therapeutic imaging assessments in 20 evaluable patients with metastatic renal cell cancer (RCC) and an early post therapy assessment at baseline and at various early time points (1 week in 5 patients, 2 weeks in 5 patients, 3 weeks in 5 patients and 4 weeks in 5 patients) after institution of standard approved sunitinib therapy at 37.5 mg/day. The clinical imaging biomarkers will include an assessment of tumor metabolism [Bannasch 1986, Frauwirth 2002, Garber 2006, Kelloff 2005, Pauwels 1998, Semenza 2001, Smith 1999, Smith 2000, Sokoloff 1977, Warburg 1956, Weber 1977A, Weber 1977B] (dynamic FDG-PET); tumor proliferation [Rasey 2002,Shields 2001, Shields 1998, Vesselle 2002, Schwartz 2003] (dynamic FLT-PET); tumor blood flow (H215O-PET, DCE MRI)[Lodge 2000], tumor perfusion (DCE-MRI)[Tofts 1999, Tofts 1997, Parker 1999]; and tumor blood volume (H215O-PET, DCE MRI)[Lodge 2000, Tofts 1999, Tofts 1997] in the same patient at baseline and then in the same patient at one of the post therapy time points (1 week, 2 weeks, 3 weeks or 4 weeks). We hypothesize that by using this set of imaging assessments it will be possible to determine an individual or more likely a set of imaging derived biomarkers that will accomplish several of the goals of the initiative which is providing funding for the study.

DETAILED DESCRIPTION:
Our proposed clinical study will:

* Provide an exploratory yet reliable and validated cadre of imaging studies done in patients that yield a mechanistically-based understanding of: 1) predictive assays for clinical benefit from standard sunitinib therapy, 2) measurement of efficacy during standard sunitinib therapy, and 3) prognosis or other long term outcomes.
* Reveal a more detailed understanding of the in vivo mechanism of standard sunitinib therapy in patient tumors, mechanistic information on why particular functional imaging patterns are seen in treated patients, and clinical measures that are useful to physicians for decision making and for explanation of efficacy or outcomes for patients.
* Predict which patients may benefit from standard sunitinib therapy.
* Determine early in the course of treatment whether standard sunitinib therapy will be efficacious and whether this can be used in future comparable patients.
* Show the outcome of patients with standard sunitinib treatment.
* Shed further information on the biological mechanism for the rapid decrease of FDG uptake on FDG-PET imaging with standard sunitinib treatment.

It is our hypothesis that a set of biologically relevant imaging biomarkers (tumor metabolism assessed with dynamic FDG-PET; tumor proliferation assessed with dynamic FLT-PET; tumor blood flow assessed with H215O-PET and DCE MRI); tumor perfusion assessed with DCE-MRI; and tumor blood volume/volume of distribution assessed with H215O-PET and DCE MRI) in the same patient at baseline and then in the same patient at one of the post therapy time points (1 week, 2 weeks, 3 weeks or 4 weeks) will provide either alone or more likely in combination information that will predict which patients will most likely benefit from standard sunitinib therapy and that an early response assessment is possible that is predictive of a durable response to the therapeutic drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older for inclusion in this study. Since there is no experience with [F-18]FLT in children and it would be inappropriate to study individuals under the age of 18 until more safety data is available.

  * After entry into the study, patients are expected to be followed for at least 2 months as part of standard of care.
  * All patients, or their legal guardians, must sign a written informed consent and HIPAA authorization in accordance with institutional guidelines.
  * The patient, if female, must be postmenopausal for a minimum of one year or surgically sterile, or on one of the following methods of birth control for a minimum of one month prior to entry into this study: IUD, oral contraceptives, Depo-Provera or Norplant. These criteria can be waived at the discretion of the investigator if the patient's tumor is considered life threatening and the one month wait required is not in the best interest of the patient. Negative pregnancy test is accepted.
  * Pre-treatment laboratory tests for patients receiving [F-18]FLT must be performed within 21 days prior to study entry. These must be less than 4 times below or above the upper or lower limit range for the respective laboratory test. These will include liver enzymes (SGOT, SGPT, ALK Phos, GGT, LDH), bilirubin (direct and total), amylase, serum electrolytes, CBC with platelets and absolute neutrophil counts, prothrombin time, partial thromboplastin time, BUN, creatinine, and urinalysis.

    * Pre-treatment radiological clinical scans/studies (Gd- enhanced MRI or CT to document metastatic renal cell carcinoma) must be performed within 30 days of study entry.

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals or Gd used in MRI imaging. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.

  * Patients who are pregnant or lactating or who suspect they might be pregnant.
  * Adult patients who require monitored anesthesia for PET or MRI scanning.
  * HIV positive patients due to the previous toxicity noted with FLT.
  * Renal Insufficiency Exclusion for MRI contrast injection. All subjects will be screened as to their renal status and those patients with renal insufficiency will be excluded from undergoing a dynamic contrast enhanced MRI scan. This is in response to the recent association of MRI contrast agents with the development of Nephrogenic Systemic Fibrosis (NSF). The patient will have a creatinine value determined within 4 weeks prior to the proposed MRI scan and have a GFR determined from the creatinine value and other data that can be used at various websites to determine the GFR. If the GFR is greater than 60 ml/min/then the patient will be deemed eligible for contrast injection. If the GFR value is between 40 ml/min and 60 ml/min the risk versus benefit of performing the contrast injection will be discussed with the referring physician and the patient. If the GFR is less than 40 ml/min the dynamic contrast study will not be performed. The non-contrast MRI scan however will be obtained for anatomic reference for the PET studies.

MRI exclusion criteria:

* Presence of any ferromagnetic metallic implants or foreign bodies, including pacemakers and certain types of stents and orthopedic hardware.
* Claustrophobia or inability to remain stationary within MRI system for ~30-45 minutes.
* Inability to breath hold for periods of at least 20 seconds.
* Known history of adverse reaction to Gd chelate contrast agents.
* Pregnancy or breastfeeding.
* Non-imageable tumor, including tumors with smallest dimension less than 10mm or tumors located in regions excessively affected by susceptibility artifacts at bone- and air-tissue interfaces or motion artifacts due to peristalsis or pulsatile flow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Hoffman, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Horn KP, Yap JT, Agarwal N, Morton KA, Kadrmas DJ, Beardmore B, Butterfield RI, Boucher K, Hoffman JM. FDG and FLT-PET for Early measurement of response to 37.5 mg daily sunitinib therapy in metastatic renal cell carcinoma. Cancer Imaging. 2015 Sep 3;15(1):15. doi: 10.1186/s40644-015-0049-x. PMID 26335224

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Sunitinib 37.5 mg: Sunitinib: Imaging studies with complete analyses for patients prior to initiation of sunitinib therapy at 37.5 mg orally/day, and at time points between 1 and 4 weeks after initiation of sunitinib therapy.
Period: Overall Study
Arm/Group | Arm 1 - Sunitinib 37.5 mg
Started | 25
Completed | 20
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 - Sunitinib 37.5 mg
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 67 [50 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Response
Description: Number of patients achieving metabolic response (at least Partial Response) assessed with follow-up FDG-PET scans compared to baseline using the European Organization for Research and Treatment of Cancer (EORTC) response criteria based on the change in the follow-up average maximum standardized uptake value (SUVmax) relative to baseline as follows: Partial Response (PR) ≥ 25% decrease in SUVmax; Progressive Disease (PD) ≥ 25% increase in SUVmax; Stable Disease (SD) < 25% change in SUVmax.
Time Frame: 4 weeks
Population: Nineteen patients were included in the analysis. One patient was found to have pathologically proven sarcoidosis at the location of the PET imaging and was therefore removed from analysis.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Sunitinib 37.5 mg
Number analyzed (Participants) | 19
participants | 5

2. Primary Outcome: Proliferative Response
Description: Number of patients achieving proliferative response (at least Partial Response) assessed with follow-up FLT-PET scans compared to baseline using the European Organization for Research and Treatment of Cancer (EORTC) response criteria based on the change in the follow-up average SUVmax relative to baseline as follows: Partial Response (PR) ≥ 25% decrease in SUVmax; Progressive Disease (PD) ≥ 25% increase in SUVmax; Stable Disease (SD) < 25% change in SUVmax.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm 1 - Sunitinib 37.5 mg
Number analyzed (Participants) | 19
participants | 9

3. Secondary Outcome: Overall Survival
Description: The length of time from the start of treatment for a disease that patients are still alive; no time limit was imposed on data collection
Time Frame: 2399 days
Population: All patients that received study treatment and PET scans at baseline and follow-up
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1 - Sunitinib 37.5 mg
Number analyzed (Participants) | 20
days | 667.5 [27 to 2399]

ADVERSE EVENTS:
Arm/Group | Arm 1 - Sunitinib 37.5 mg
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Sunitinib 37.5 mg (N=25)
Syncope (Nervous system disorders) | 1
Infection: Urinary Tract (Renal and urinary disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Obstruction: Bowel (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Muscle Weakness - Extremity Lower (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Sunitinib 37.5 mg (N=25)
Alkaline Phosphatase: Increased (Metabolism and nutrition disorders) | 2 (2)
ALT Increase (Metabolism and nutrition disorders) | 2 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
AST Increase (Metabolism and nutrition disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine Increased (Metabolism and nutrition disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 6 (7)
Glutamyl transpeptidase: increase (Metabolism and nutrition disorders) | 3 (3)
Hemoglobin: decrease (Blood and lymphatic system disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Infection: Urinary Tract (Renal and urinary disorders) | 2 (2)
Leukocytes: decrease (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 8 (8)
Obstruction: bowel (Gastrointestinal disorders) | 2 (2)
Pain: Oral Cavity (Gastrointestinal disorders) | 2 (2)
Partial Thromboplastin Time increase (Blood and lymphatic system disorders) | 4 (4)
Platelets: decrease (Blood and lymphatic system disorders) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes